CLINICAL TRIAL: NCT04702022
Title: Non-invasive Diagnosis and Management of Subclinical Rejection in Kidney Transplant Patients Using 18F-fluorodeoxy Glucose Positron Emission Tomography (18FDG-PET/CT)
Brief Title: Added Value of 18 FDG Pet-scanner in Diagnosis and Management of Subclinical Rejection in Kidney Transplant Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Antoine Bouquegneau, Principal Investigator, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Liege AVOID
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-05

CONDITIONS: Kidney Transplant Rejection; Kidney Transplant; Complications
Keywords: PET/CT imaging; Corticoids withdrawal; SubClinical Rejection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Humoral Arm (Other): The renal biopsy shows signs of humoral rejection: the patient is excluded from the study and is treated "as usual" on the basis of the histological results.
  Interventions: Diagnostic Test: 18FDG PET / CT
- "Highly Metabolic patients" (Other): The renal biopsy does not show signs of humoral rejection but the 18FDG PET / CT shows a high metabolic activity of the graft (> 2.4): the patient is treated "as usual" on the basis of histological findings.
  Interventions: Diagnostic Test: 18FDG PET / CT
- " Low metabolic patients" (Other): The renal biopsy does not show signs of humoral rejection and the 18FDG PET / CT shows a weak metabolic activity of the graft (<2.4): the immunosuppressive treatment is gradually weaned off corticosteroids.
  Interventions: Diagnostic Test: 18FDG PET / CT

INTERVENTIONS:
Diagnostic Test: 18FDG PET / CT — The PET/CT procedure was performed using cross-calibrated Philips Gemini TF Big Bore or TF 16 PET/CT systems (Philips Medical Systems, Cleveland, OH) at 201 18 minutes following intravenous injection of a mean dose of 3.2 0.2 MBq/kg of body weight of 18 F-FDG. A low-dose helical CT (5-mm slice thickness, 120-kV tube voltage, and 40-mAs tube current-time product) centered to the renal transplant was performed, followed by PET scanning with two bed positions, each lasting 240 seconds. Images were reconstructed using iterative list mode time-of-flight algorithms. Corrections for attenuation, dead time and random and scatter events will be applied.

SUMMARY:
The renal biopsy (RB) represents the gold-standard for the diagnosis of acute renal transplant rejection (AR), and allows early verification of a so-called "subclinical" rejection, ie without any clinical or biological abnormality detectable in a stable kidney transplant patient. The RB also makes it possible to certify a strictly normal renal histology and thus to motivate the withdrawal of corticosteroid therapy. It is this 3-month post-transplant protocol RB protocol that has been effective since 2007 at the CHU Liège.

However, RB is an invasive procedure, contraindicated in patients taking anticoagulants, and carrying a significant risk of complications. The potential complications associated with RB motivate the identification and validation of other diagnostic means. In the present project, the investigators propose to study the relevance of positron emission tomography (PET), coupled with conventional tomography (CT), after intravenous injection of 18-fluoro-deoxy-glucose (18FDG) in the overall protocol of the renal transplant patient at 3 months post-transplant to:

(i) allow protocol renal biopsy only in patients with suspicion of an acute rejection (ii) be a decision maker for withdrawal from corticosteroids in the absence of rejection

In practice, the investigators suggest performing 18FDG PET / CT imaging on the day of the surveillance biopsy, which is systematically performed in all kidney transplant patients at University Hospital of Liège 3 months after transplant. The investigators are considering 3 scenarios:

* Scenario 1. The renal biopsy shows signs of humoral rejection: the patient is excluded from the study and is treated "as usual" on the basis of the histological results.
* Scenario 2. The renal biopsy does not show signs of humoral rejection but the 18FDG PET / CT shows a high metabolic activity of the graft (> 2.4): the patient is treated "as usual" on the basis of histological findings.
* Scenario 3. The renal biopsy does not show signs of humoral rejection and the 18FDG PET / CT shows a weak metabolic activity of the graft (<2.4): the immunosuppressive treatment is gradually weaned off corticosteroids.

This clinical research project is interested in a major health problem in the follow-up of renal transplant patients, and could make it possible to improve the management of a subclinical rejection of the renal transplant and to increase the withdrawal of corticosteroids including side effects are well known.

DETAILED DESCRIPTION:
Subclinical rejection (SCR) has been defined as "the documentation by light histology of unexpected evidence of acute rejection (AR) in a stable patient". The diagnosis of SCR is important given that the treatment of subclinical T-cell-mediated AR results in similar long-term graft survival to that in patients without rejection. Surveillance transplant biopsies are, by definition, required for the diagnosis of SCR. Still, only 17% of transplant centers in the United States perform surveillance biopsies in all patients, whereas 62% do not perform surveillance biopsies at all because the incidence of SCR is low3. Non-invasive biomarkers may thus be developed as "rule out" tests, with the highest negative predictive value, in order to reduce the indiscriminate use of allograft biopsies in stable kidney transplant recipients (KTR). Beside urine-derived and blood-based biomarkers of SCR, the investigators have recently reported in a monocentric prospective pilot study that 18F-Fluorodeoxyglucose Positron Emission Tomography coupled with Computed Tomography (18F-FDG PET/CT) non-invasively rules out SCR at ~3 months post kidney transplantation (KTx).

In previous 92-patient cohort published by the investigators, the ratio between the mean standardized 18F-FDG uptake values (SUVs) of the renal allograft and the psoas muscle (used as reference tissue) was significantly higher in the group with biopsy-proven SCR versus the group with strictly normal histology. The area under the ROC curve (AUC) reached 0.79, with a negative predictive value of 98% using an mSUVR threshold of 2.4.

All adult KTR who undergo surveillance transplant biopsy at ~3 months post KTx are eligible for the present study, except pregnant women and patients PCR-proven BK nephropathy. Written informed consent will be obtained. KTx will be performed in accordance with the Declaration of Istanbul. Surveillance biopsies will be locally (in each participating centers) and centrally (at ULiège CHU) assessed by pathologists blinded to the results of 18F-FDG PET/CT. Banff 2017 classification will be conventionally used. Total inflammation (ti) will take into account interstitial inflammation in both non-sclerotic and sclerotic areas. C4d staining will be performed in all cases. PET/CT will be performed with late acquisitions (~180 minutes) after 18F-FDG intravenous injection (~3 Mbq/kg) within a 48-hour period around the biopsy, before any modification of immunosuppressive regimens. The mean standardized uptake value (mSUV) of kidney cortex will be measured and averaged from 4 volumes of interest (VOI) distributed in the upper (n=2) and lower (n=2) poles, both locally (in each participating centers) and centrally (at ULiège CHU)10. The mSUV of kidney will be normalized to the mSUV of psoas muscle (VOI of 20 ml) or the liver (VOI of 20 ml), considered as reference tissues in order to obtain the corresponding mean SUV Ratios (mSUVR).

The patients will be afterwards in one of these three categories :

1. The renal biopsy shows signs of humoral rejection: the patient is excluded from the study and is treated "as usual" on the basis of the histological results.
2. The renal biopsy does not show signs of humoral rejection but the 18FDG PET / CT shows a high metabolic activity of the graft (> 2.4): the patient is treated "as usual" on the basis of histological findings.
3. The renal biopsy does not show signs of humoral rejection and the 18FDG PET / CT shows a weak metabolic activity of the graft (<2.4): the immunosuppressive treatment is gradually weaned off corticosteroids.

The goals are :

(i) to use the measurement of renal accumulation of the 18FDG marker at the level of the renal graft as a non-invasive indicator of the absence of a subclinical cellular rejection and to use the information from the renal biopsy only if the metabolic activity of the graft is increased.

(ii) to use the measurement of renal accumulation of the 18FDG marker in the renal graft as a non-invasive indicator of the absence of cell rejection and to initiate the withdrawal of corticosteroids if the metabolic activity of the graft is normal.

ELIGIBILITY:
Inclusion Criteria:

* Kidney recipients aged over 18 and of all sexes

Exclusion Criteria:

* Pregnant patients
* Polyomavirus nephropathy
* Highly sensitised patients (historical or at 3 months Donor specific antibodies)
* No corticosteroids withdrawal allowed (second kidney transplantation or primary disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of rejection with 18 FDG data | at 3 months
  use the measurement of renal accumulation of the 18FDG marker at the level of the renal graft as a non-invasive indicator of the absence of a subclinical cellular rejection and to use the information from the renal biopsy only if the metabolic activity of the graft is increased.
Withdrawal of corticosteroids with 18FDG data | At 6 months
  use the measurement of renal accumulation of the 18FDG marker in the renal graft as a non-invasive indicator of the absence of cell rejection and to initiate the withdrawal of corticosteroids if the metabolic activity of the graft is normal

SECONDARY OUTCOMES:
Allograft rejection | at 6 months and 1year
  Incidence of rejection in patient with corticosteroids withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Francois Jouret, Principal Investigator — University of Liege
Locations (1):
- Antoine Bouquegneau, Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No